CLINICAL TRIAL: NCT01588262
Title: Early Rehabilitation of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Uppsala University (Other); University of Agder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REKnr 2010/1911
Record Dates: First submitted 2012-01-30; First posted 2012-04-30 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2015-10

CONDITIONS: Breast Cancer; Colorectal Cancer; Lymphoma; Prostate Cancer; Testicle Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lymphoma; Prostatic Neoplasms; Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stressmanagement counselling (Other)
  Interventions: Other: Stressmanagement
- Control (No Intervention)

INTERVENTIONS:
Other: Stressmanagement — Individual stepped-care approach stressmanagement by specially trained counsellor
  Other Names: I-a; I-b
  Arms: Stressmanagement counselling

SUMMARY:
A life threatening disease such as cancer may lead to post traumatic stress disorder, and even when reporting low levels of side-effects from cancer disease and treatment, 80% report high levels of stress symptoms. The purpose of the present randomised controlled trial is to examine the psychosocial effects of a stress management intervention based on cognitive behaviour therapy and with focus on increased physical activity in patients with various cancer diagnoses using a stepped-care approach. When using a stepped-care approach it is possible to study the level and intensity of stress management intervention required to achieve increased well-being. A cost-utility analysis will also be performed. 300 adult patients with a recent diagnosis of breast-, colorectal- prostate, testicular cancer or lymphoma and scheduled for adjuvant and/or curative oncologic treatment at Haukeland University Hospital, will be consecutively included in the prospective intervention study. The patients will be randomized to intervention or control. In step 1, all patients in the intervention group (I-a) will receive 2 counselling sessions. Patients who report clinically significant levels of stress, such as intrusive thoughts/avoidance behaviour (measured by Impact of Event Scale) and/or worry and depressions (measured by Hospital and Depression Scale) will be included in Step 2 (I-b) and include another 4-7 counselling sessions. There will also be a focus on motivating to increase physical activity level. Both the intervention (I) and control group (C) are allowed to take part in the common rehabilitation program with patient education and physical training. Data will be collected with self-reported standardized questionnaires. Objectively measures of physical activity level, sleep and daily energy expenditure are recorded with SenseWear™ Pro3 Armband. Measure point is at inclusion and than after 6 week, 4, 8, 12 and 24 month.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with breast cancer,
* colorectal cancer,
* lymphoma,
* prostate cancer or testicle cancer and scheduled for adjuvant and/or curative treatment in the form of chemotherapy, radiation therapy and/or hormonal therapy at the Department of Oncology and Medical physics, Haukeland University Hospital, (Dept. of Oncology) Bergen,
* residence in Rogaland, Hordaland and Sogn and fjordane county council,
* initial treatment for cancer

Exclusion Criteria:

* An ongoing psychiatric condition,
* language deficiencies in Norwegian,
* surgery for prostate cancer (only applies for prostate cancer) patients),
* men with breast cancer,
* live in nursing homes,
* previous cancer,
* treated for cancer earlier,
* already implemented oncological treatment,
* not self-reliant

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in psychosocial status | from baseline to 24 month

SECONDARY OUTCOMES:
Cost effectiveness of the stress-management intervention. | 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology and Medical Physics, Cancer center for Education and rehabilitation, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Arving C, Thormodsen I, Brekke G, Mella O, Berntsen S, Nordin K. Early rehabilitation of cancer patients - a randomized controlled intervention study. BMC Cancer. 2013 Jan 7;13:9. doi: 10.1186/1471-2407-13-9. PMID 23294513